CLINICAL TRIAL: NCT02353494
Title: Efficacy and Safety of Dihydroartemisinin-piperaquine for the Treatment of Uncomplicated Plasmodium Falciparum and Plasmodium Vivax Malaria in Timika, Indonesia
Brief Title: Efficacy and Safety of Dihydroartemisinin-piperaquine (DHP) for the Treatment of Uncomplicated Malaria
Status: Completed | Type: Observational
Sponsor: Menzies School of Health Research (Other)
Collaborators: Eijkman Institute for Molecular Biology (Other); World Health Organization (Other)
Responsible Party: Sponsor
Other Study IDs: Indonesia DHP 2013
Record Dates: First submitted 2015-01-28; First posted 2015-02-02 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Plasmodium Falciparum Infection; Plasmodium Vivax Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples for genotyping of Plasmodium vivax and Plasmodium falciparum.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Dihydroartemisinin-Piperaquine — Treatment according to national guidelines with follow up.

SUMMARY:
This is an observational safety and efficacy study on dihydroartemisinin-piperaquine in Timika, Indonesia with a 42 day follow up period.

DETAILED DESCRIPTION:
Dihydroartemisinin-piperaquine (DHA-Pip) is part of the current national guidelines for the treatment of uncomplicated malaria in Indonesia. In order to guarantee safe and efficacious treatment for all patients diagnosed with uncomplicated malaria in the area, it is essential to monitor the effectiveness of the recommended treatment from a clinical perspective and assess whether the provided treatment is safe for recipients. This trial re-evaluates the local efficacy and safety of DHA-Pip for P. falciparum and P. vivax infections.

Patients with uncomplicated malaria attending a public health care facility in Timika, Papua, Indonesia, who meet the study inclusion criteria will be enrolled, treated on site with DHA-Pip and followed up for 42 days. The follow-up will consist of a fixed schedule of check-up visits and corresponding clinical and laboratory examinations. On the basis of the results of these assessments, the patients will be classified as having therapeutic failure (early or late) or an adequate response. The proportion of patients experiencing therapeutic failure and drug related adverse events during the follow-up period will be used to estimate the efficacy and safety of the study drug. PCR analysis will be used to distinguish between a true recrudescence due to treatment failure and episodes of reinfection.

The outcome of the proposed project will have a direct impact on the decision making process of the Indonesian Ministry of Health on whether there is a need to alter the existing antimalarial treatment guidelines.

ELIGIBILITY:
Inclusion criteria:

* age between one year (weight more than 5 kgs) to 65 years old;
* mono-infection with Plasmodium falciparum or Plasmodium vivax detected by microscopy;
* parasitaemia of more than 1000/μl asexual parasites for P. falciparum and more than 250/μl asexual parasites for P. vivax
* presence of axillary temperature ≥ 37.5 °C or history of fever during the past 24 h;
* ability to swallow oral medication;
* ability and willingness to comply with the study protocol for the duration of the study and to comply with the study visit schedule; and
* informed consent from the patient or from a parent or guardian in the case of children.

Exclusion criteria:

* presence of general danger signs in children aged under 5 years or signs of severe falciparum malaria according to the definitions of WHO
* mixed or mono-infection with another Plasmodium species detected by microscopy;
* presence of severe malnutrition (defined as a child whose growth standard is below -3 z-score, has symmetrical oedema involving at least the feet or has a mid-upper arm circumference < 110 mm);
* presence of febrile conditions due to diseases other than malaria (e.g. measles, acute lower respiratory tract infection, severe diarrhoea with dehydration) or other known underlying chronic or severe diseases (e.g. cardiac, renal and hepatic diseases, HIV/AIDS);
* regular medication, which may interfere with antimalarial pharmacokinetics;
* history of hypersensitivity reactions or contraindications to dihydroartemisinin-piperaquine
* a positive pregnancy test or breastfeeding

Ages: 12 Months to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients suffering from uncomplicated Plasmodium falciparum / Plasmodium vivax infections attending the study hospital during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2015-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
The proportion of adverse and serious adverse observed during the follow up period | 6 months
The cumulative incidence of success and failure rates at day 42, PCR-uncorrected and PCR-corrected | 6 months

SECONDARY OUTCOMES:
Proportion of patients aparasitaemic on days 1 and 2 | 6 months
Haematological recovery | 6 months
Gametocyte carriage during follow up | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne R Poespoprodjo, MD, PhD, Principal Investigator — Timika Research Facility Kompleks RSMM, Timika-Papua, Indonesia
Locations (1):
- Timika District Hospital, Timika, Indonesia